CLINICAL TRIAL: NCT02717000
Title: Non-invasive Diagnosis of Non-alcoholic Steatohepatitis in Patients With Non-alcoholic Fatty Liver Disease Using Markers and Imaging Techniques
Brief Title: NASH: Non-invasive Diagnostic Markers and Imaging
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Zuyderland Medical Centre (Other)
Responsible Party: Principal Investigator, Ger Koek, MD, PhD, Maastricht University Medical Center
Other Study IDs: 15-T-167
Record Dates: First submitted 2016-03-15; First posted 2016-03-23 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Nonalcoholic Fatty Liver Disease; Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, exhaled air, feces

GROUPS / COHORTS (2):
- NASH
- No NASH

SUMMARY:
Rationale:

Non-alcoholic fatty liver disease (NAFLD) is the most widespread liver disorder in Western society (prevalence 20-30%). It is strongly associated with overweight and obesity. The majority of patients have simple steatosis. However, in about 15-30% of the subjects, a chronic inflammatory state develops that is referred to as non-alcoholic steatohepatitis (NASH), which leads to an overall increase in morbidity and mortality due to the progression to fibrosis, cirrhosis and in some cases, hepatocellular carcinoma (HCC). The term NAFLD comprises both simple steatosis and NASH. Most patients with NAFLD have no or few, mainly aspecific symptoms; and generally there is a silent progression of simple steatosis to NASH and in the end, liver-related morbidity and mortality.

To date, liver biopsy is the most sensitive test for detecting and staging NAFLD, and is the only reliable method for differentiating between NASH and simple steatosis. However, the procedure of obtaining a liver biopsy is invasive and associated with patient discomfort, significant complications and high costs. In addition, liver biopsy is prone to sampling error and inter- and intra-observer variability, due to the small size of liver biopsy samples. This method is therefore not suitable for screening large numbers of subjects at risk, or for follow-up of patients with NASH over time. Hence, only subjects at high risk (usually based upon elevated aminotransferase levels, which is not specific for the presence of NASH) are biopsied, leading to an underestimation of NASH prevalence and undertreatment. Further insight into disease mechanisms and risk factors for NAFLD and in particular NASH is warranted, to enable early diagnosis, adequate therapy and preventive measures to improve health status of these individuals. Accurate and less invasive methods to evaluate NASH, and NAFLD, are urgently needed.

Objective: The primary objective of this study is to establish non-invasive tools (e.g. biomarkers and imaging) to accurately diagnose patients with NASH. The secondary objective is to show an association between the levels of identified markers and disease severity.

Study design:

Eligible subjects will be included via the outpatient clinics Zuyderland in Heerlen, the Catharina hospital in Eindhoven and MUMC+ in Maastricht. A subset of eligible subjects has undergone a liver biopsy for clinical reasons. It is estimated that about 85% of subjects will be asked to undergo a biopsy for study purposes only. Liver biopsies for study purposes will be performed during a surgical procedure, e.g. bariatric surgery or cholecystectomy.

Blood, faeces and exhaled air will be collected and a FibroScan (+CAP) will be performed during a study visit. An MRI will be performed, to estimate the degree of steatosis. Furthermore, anthropometric data (weight, height, abdominal and waist circumference and blood pressure (BP)) will be collected.

The participants in the group undergoing liver biopsy during bariatric surgery will be asked permission to be approached for follow-up measurements 3 months post-surgery. As they will lose weight, which is associated with improvement of hepatic steatosis, this enables assessment of possible changes over time. A routine follow-up visit post-surgery will take place after 3 months. The follow-up measurements will be combined with this visit, minimizing the burden for the participant. The measurements will consist of blood, faeces and exhaled air collection and a FibroScan (+CAP) will be performed during a study visit. Furthermore, weight, height, BP and abdominal and waist circumference will be measured.

Study population:

Subjects with proven NAFLD by histology or NAFLD proven by imaging, who are undergoing surgery (i.e. bariatric surgery or cholecystectomy) will be asked to participate in this study. Furthermore, all subjects have to be between 18 and 65 years old.

Main study parameters/endpoints:

Non-invasive tool based on biomarkers and imaging to diagnose NASH.

ELIGIBILITY:
Inclusion Criteria:

* NAFLD proven by imaging
* Age 18-65 years

Exclusion Criteria:

* Incompetent to understand and/or sign the informed consent.
* Ethanol consumption exceeding more than 14 standard beverages per week for males and more than 7 standard beverages per week for female.
* Causes for secondary hepatic fat accumulation such as significant alcohol consumption, medications, Wilson's disease, viral infections, starvation or parenteral nutrition, among others, and conditions associated with microvesicular steatosis
* Not willing to be informed about unexpected findings by MRI and histopathologic evaluation of liver biopsy
* Unwilling to collect biosamples.
* Pregnancy and breastfeeding.
* Diagnosis of liver cirrhosis and/or hepatocellular carcinoma.
* Current diagnosis of extrahepatic malignancie(s) or prior diagnosis within last 5 years.
* Diagnosis of chronic inflammatory disease (i.e. inflammatory bowel disease, rheumatoid arthritis, inflammatory lung disease, severe infectious diseases), other than NAFLD/NASH
* Chronic use of immunosuppressants (e.g. biologicals, prednisolone, azathioprine)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with proven NAFLD by histology or NAFLD proven by imaging, who are undergoing surgery (i.e. bariatric surgery or cholecystectomy) will be asked to participate in this study. Furthermore, all subjects have to be between 18 and 65 years old.
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Non-invasive tool to diagnose NASH (based on imaging (TE/MRI) an markers (biochemical, volatile organic compounds) | once enough evaluable patients are recruited, an average of 1 year